CLINICAL TRIAL: NCT06545045
Title: Pilot Testing of Metacognitive Strategy Training to Address Cancer-related Cognitive Impairment in Breast Cancer
Brief Title: Cognitive Rehabilitation Following Breast Cancer Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anna Boone, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2101565; 1R21CA286404 (NIH)
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Female
Keywords: Cancer; Breast Cancer; Cognition; Metacognition; Activities of daily living
MeSH Terms: conditions — Neoplasms; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All outcomes assessors will be blinded to participant study group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metacognitive strategy training (MCST) (Experimental): Each MCST session will be follow the procedures of Cognitive Orientation to daily Occupational Performance (CO-OP) intervention. There will be 10, 45-minute, weekly sessions. All sessions will be delivered in-person with a trained occupational therapist.
  Interventions: Behavioral: Metacognitive Strategy Training (MCST)
- Inactive Control Group (Active Comparator): Participants will receive a weekly phone call from study staff to maintain contact and monitor changes in activity.
  Interventions: Behavioral: Inactive Control Group

INTERVENTIONS:
Behavioral: Metacognitive Strategy Training (MCST) — The MCST group will follow procedures for the Cognitive Orientation to daily Occupational Performance intervention. First, five functional, everyday life goals are identified collaboratively by the participant and interventionist. In the second meeting, the therapist introduces the approach to the subject and teach a global cognitive strategy (i.e., GOAL-PLAN-DO-CHECK). In all subsequent sessions, this strategy is used as the main problem-solving framework to facilitate skill acquisition. The subject identifies a GOAL, and then is guided by the therapist to discover a PLAN to potentially achieve the goal. The subject is then asked to DO the plan (if feasible during the therapy session otherwise asked to complete at home prior to the next treatment session), and subsequently to CHECK to see if the plan worked, i.e. the goal was achieved. This process is repeated until satisfactory performance is met for each established goal.
  Arms: Metacognitive strategy training (MCST)
Behavioral: Inactive Control Group — Weekly contact will be made via telephone call to (1) maintain study engagement, (2) introduce weekly social contact with researchers, mimicking some of the potential incidental effects of the experimental group, and (3) ascertain what, if any, additional steps participants have taken to reduce cognitive symptoms. The content of each of these meetings will be tracked in intervention notes.
  Arms: Inactive Control Group

SUMMARY:
The goal of this proposed project is to evaluate the feasibility and preliminary effect of metacognitive strategy training to improve activity performance, cognition, and quality of life in breast cancer survivors with cancer-related cognitive impairment (CRCI). The other goal of this proposed project is to examine the effects of CO-OP on resting (rsFC)- and task-state functional connectivity as compared to an inactive control group.

DETAILED DESCRIPTION:
Breast cancer survivors often self-report cognitive deficits, primarily in executive functioning (planning, problem solving, multitasking), memory, and processing speed after cancer treatment, i.e., cancer-related cognitive impairment (CRCI). The prevalence of CRCI following breast cancer is as high as 78% and can persist chronically after treatment has ended. In other health conditions associated with cognitive impairment, such as traumatic brain injury, the only evidence-based recommended practice standard for deficits in executive function is metacognitive strategy training (MCST). In this approach, participants are taught a general cognitive strategy that can be applied in known and novel contexts to devise task specific strategies to successfully engage in an activity. While the cognitive deficits identified in and described by breast cancer survivors seem quite amenable to MCST, there is no study in the published literature which measures the efficacy of MCST on CRCI. The Cognitive Orientation to daily Occupational Performance (CO-OP) approach is a MCST intervention in which subjects are taught a general cognitive strategy that can be applied in known and novel contexts to devise task specific strategies to engage in an activity. Preliminary data suggest that CO-OP may have a positive impact on subjective and objective cognitive performance in breast cancer survivors with CRCI. Further, this study will evaluate the neurophysiological underpinnings associated with treatment changes through the use of neuroimaging methods.

ELIGIBILITY:
Inclusion Criteria:

* self-reported CRCI (Global Rating of Cognition dysfunction as "Moderately" "Strongly "or "Extremely" AND a Cognitive Failures Questionnaire1 (CFQ) score >30)
* completed treatment for active cancer diagnosis (invasive ductal or lobular BrCA Stages I, II, or III) at least 6 months but not greater than 3 years prior to participation
* able to read, write, and speak English fluently
* able to provide valid informed consent
* have a life expectancy of greater than 6 months at time of enrollment
* on stable doses (i.e., no changes in past 90 days) of medications that are known to impact cognitive function (i.e., anti-depressants)

Exclusion Criteria:

* prior cancer diagnoses of other sites with evidence of active disease within the past year
* active diagnoses of any acute or chronic brain-related neurological conditions that can alter normal brain anatomy or function (e.g., Parkinson's disease, dementia, cerebral infarcts) dementia symptoms as indicated by a score of <23 on the Montreal Cognitive Assessment (MoCA)
* severe depressive symptoms (Personal Health Questionnaire-9 (PHQ-9) score of ≥21)
* history of severe traumatic brain injury, prolonged loss of consciousness (e.g., coma)
* conditions contraindicated for MRI (e.g., electrical implants, pumps, claustrophobia)
* blue-yellow colorblindness
* pregnancy

The screening methods identified in parentheses next to appropriate inclusion/exclusion criteria will be used to verify appropriate selection of study participants.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility measures | After study completion, an average of 12 weeks
  Recruitment rate, retention rate
Canadian Occupational Performance Measure (COPM) Performance | Pre-intervention (week 0) and post-intervention (week 12)
  Self-report measure of activity performance. Minimum = 1, Maximum = 10. Higher scores mean better performance.
Canadian Occupational Performance Measure (COPM) Satisfaction | Pre-intervention (week 0) and post-intervention (week 12)
  Self-report measure of activity performance. Minimum = 1, Maximum = 10. Higher scores mean better performance.

SECONDARY OUTCOMES:
Cognitive Failures Questionnaire (CFQ) | Pre-intervention (week 0) and post-intervention (week 12)
  Self-report measure of lapses in motor function memory and perception. This questionnaire contains 25 items and scores range from 0 to 100. Higher scores = greater perceived impairment.
Dysexecutive Questionnaire (DEX) | Pre-intervention (week 0) and post-intervention (week 12)
  Self-report measure of the functional impact of executive dysfunction. It consists of 20 items within four domains: (1) emotional, (2) motivational, (3) behavioral, and (4) cognitive. Each item is rated for frequency using a 5-point Likert scale ranging from 0 (never) to 4 (very often).
Trail Making Test (TMT) | Pre-intervention (week 0) and post-intervention (week 12)
  Part A is an attention, visual search, and motor speed task that involves connecting a series of numbers in ascending order. Part B requires alternating between numbers and letters to assess set shifting and executive abilities.
Controlled Oral Word Association (COWA) | Pre-intervention (week 0) and post-intervention (week 12)
  Measure of verbal fluency that requires spontaneous word production for a different letter of the alphabet across three different trials.
The Activity Card Sort (ACS) | Pre-intervention (week 0) and post-intervention (week 12)
  Self-report measure of participation in various everyday life activities that are in the categories of low demand leisure, high demand leisure, instrumental activities of daily living, and social activity. Cards are sorted according to if the subject is performing each activity as much, less than, or more as compared to before experiencing cancer-related cognitive impairment.
Functional Assessment of Cancer Therapy-Breast (FACT-B) | Pre-intervention (week 0) and post-intervention (week 12)
  A quality-of-life measure across five domains: Physical, social, emotional, functional well-being, and breast-cancer subscale.
Participation Strategies Self Efficacy Scale (PS-SES) | Pre-intervention (week 0) and post-intervention (week 12)
  Self-report measure of self-efficacy in using participation strategies. The subject rates confidence across 35 items within six subscales: (1) managing home participation, (2) staying organized, (3) planning and managing community participation, (4) managing work and productivity), (5) managing communication, and (6) advocating for resources.
Paced Auditory Serial Addition Test (PASAT) | Pre-intervention (week 0) and post-intervention (week 12)
  Measure of working memory and attention in which a series of single digit numbers are presented audibly individuals. The most recent two digits are to be summed prior to the next digit presented. Two commonly used subversions use a 2 second or 3 second inter-stimulus interval.
Hopkins Verbal Learning Test-Revised (HVLT-R) | Pre-intervention (week 0) and post-intervention (week 12)
  Measure of verbal learning and memory in which a list of 12 words is to be recalled. Three learning trials with free recall followed by a delayed recall at 20 minutes and a recognition trial.

CONTACTS AND LOCATIONS:
Overall Officials: Anna E Boone, PhD, OTR/L, Principal Investigator — University of Missouri Occupational Therapy
Locations (1):
- University of Missouri, Columbia, Missouri, United States

REFERENCES:
- [Background] Hutchinson AD, Hosking JR, Kichenadasse G, Mattiske JK, Wilson C. Objective and subjective cognitive impairment following chemotherapy for cancer: a systematic review. Cancer Treat Rev. 2012 Nov;38(7):926-34. doi: 10.1016/j.ctrv.2012.05.002. Epub 2012 Jun 2. PMID 22658913
- [Background] O'Farrell E, MacKenzie J, Collins B. Clearing the air: a review of our current understanding of "chemo fog". Curr Oncol Rep. 2013 Jun;15(3):260-9. doi: 10.1007/s11912-013-0307-7. PMID 23483375
- [Background] Schagen SB, Wefel JS. Chemotherapy-related changes in cognitive functioning. EJC Suppl. 2013 Sep;11(2):225-32. doi: 10.1016/j.ejcsup.2013.07.007. No abstract available. PMID 26217131
- [Background] Myers JS. Chemotherapy-related cognitive impairment. Clin J Oncol Nurs. 2009 Aug;13(4):413-21. doi: 10.1188/09.CJON.413-421. PMID 19648097
- [Background] Janelsins MC, Kohli S, Mohile SG, Usuki K, Ahles TA, Morrow GR. An update on cancer- and chemotherapy-related cognitive dysfunction: current status. Semin Oncol. 2011 Jun;38(3):431-8. doi: 10.1053/j.seminoncol.2011.03.014. PMID 21600374
- [Background] Wefel JS, Schagen SB. Chemotherapy-related cognitive dysfunction. Curr Neurol Neurosci Rep. 2012 Jun;12(3):267-75. doi: 10.1007/s11910-012-0264-9. PMID 22453825
- [Background] Janelsins MC, Kesler SR, Ahles TA, Morrow GR. Prevalence, mechanisms, and management of cancer-related cognitive impairment. Int Rev Psychiatry. 2014 Feb;26(1):102-13. doi: 10.3109/09540261.2013.864260. PMID 24716504
- [Background] Cicerone KD, Dahlberg C, Kalmar K, Langenbahn DM, Malec JF, Bergquist TF, Felicetti T, Giacino JT, Harley JP, Harrington DE, Herzog J, Kneipp S, Laatsch L, Morse PA. Evidence-based cognitive rehabilitation: recommendations for clinical practice. Arch Phys Med Rehabil. 2000 Dec;81(12):1596-615. doi: 10.1053/apmr.2000.19240. PMID 11128897
- [Background] Cicerone KD, Langenbahn DM, Braden C, Malec JF, Kalmar K, Fraas M, Felicetti T, Laatsch L, Harley JP, Bergquist T, Azulay J, Cantor J, Ashman T. Evidence-based cognitive rehabilitation: updated review of the literature from 2003 through 2008. Arch Phys Med Rehabil. 2011 Apr;92(4):519-30. doi: 10.1016/j.apmr.2010.11.015. PMID 21440699
- [Background] Haskins E. Cognitive Rehabilitation Manual: Translating Evidence-Based Recommendations into Practice. vol 1. American Congress of Rehabilitation Medicine; 2012.
- [Background] Wolf TJ, Doherty M, Kallogjeri D, Coalson RS, Nicklaus J, Ma CX, Schlaggar BL, Piccirillo J. The Feasibility of Using Metacognitive Strategy Training to Improve Cognitive Performance and Neural Connectivity in Women with Chemotherapy-Induced Cognitive Impairment. Oncology. 2016;91(3):143-52. doi: 10.1159/000447744. Epub 2016 Jul 23. PMID 27449501